CLINICAL TRIAL: NCT03546257
Title: Magnifying Endoscopy With Narrow Band Imaging Versus Endoscopic Ultrasonography for Prediction of Tumor Invasion Depth in Early Gastric Cancer: A Prospective Comparative Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2018-0220
Record Dates: First submitted 2018-05-21; First posted 2018-06-06 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Early Gastric Cancer; Gastric Adenoma; Gastric Dysplasia
Keywords: Early gastric cancer; Invasion depth; Narrow band imaging; Endoscopic ultrasonography
MeSH Terms: conditions — Stomach Neoplasms | interventions — Narrow Band Imaging

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EUS: group using conventional WLE and EUS
- ME-NBI: group using WLE and ME-NBI.
  Interventions: Device: magnifying endoscopy with narrow band imaging (ME-NBI)

INTERVENTIONS:
Device: magnifying endoscopy with narrow band imaging (ME-NBI) — A system consisting of a magnifying endoscope combined with narrow-band imaging (NBI), with the spectral band width narrowed by optical filters, was developed to enhance visualization of mucosal surface structure and vascular architecture. There were some reports that the magnifying endoscopy with narrow band imaging (ME-NBI) is superior to predict the histologic differentiation, depth of invasion and lesion margin than WLE.
  Groups: ME-NBI

SUMMARY:
The treatment of early gastric cancer can be divided into endoscopic resection and surgery, and the precise staging of early gastric cancer is very important to prevent unnecessary surgery or additional surgery after the procedure. The possibility of endoscopic resection is determined by the risk of lymph node metastasis. The risk factors of lymph node metastasis of early gastric cancer are lesion size, presence of ulceration, histologic differentiation, and depth of invasion. In contrast to other factors, the factor of invasion depth is relatively difficult to predict by using the conventional white light endoscopy (WLE). Therefore, the endoscopic ultrasonography (EUS) has been tried to use for prediction of the invasion depth. However, many studies reported that the accuracy of endoscopic ultrasonography for predicting the depth of invasion was varied.

A system consisting of a magnifying endoscope combined with narrow-band imaging (NBI), with the spectral band width narrowed by optical filters, was developed to enhance visualization of mucosal surface structure and vascular architecture. There were some reports that the magnifying endoscopy with narrow band imaging (ME-NBI) is superior to predict the histologic differentiation, depth of invasion and lesion margin than WLE.

In this study, we divide the patients with suspected early gastric cancer (EGC) into the two groups as group using conventional WLE and EUS and group using WLE and ME-NBI, and try to compare the accuracy of EUS and ME-NBI for predicting the invasion depth of EGC. We also try to analyze the factors that affect the accuracy for predicting of depth such as characteristics of cancer lesion and histologic differentiation of cancer in each group. In addition, we try to analyze the characteristic imaging findings of ME-NBI for early gastric cancer and gastric adenoma and evaluate the efficacy of ME-NBI for early gastric cancer and gastric adenoma diagnosis.

DETAILED DESCRIPTION:
The subjects is divided into early gastric cancer patients and gastric adenoma patients according to histologic biopsy result and white light endoscopic findings. Study 1 applies for early gastric cancer patients, Study 2 applies for gastric adenoma patients.

A) Study 1 The NBI group performs ME-NBI first before EUS. The endoscopist evaluates NBI findings such as the invasion depth and describes ME-NBI impression. And then, EUS is performed likewise. The final treatment plan is determined by the EUS result, so group assignment does not affect the final treatment plan.

The EUS group performs EUS first before NBI. The endoscopist evaluates EUS findings such as the invasion depth and describes EUS impression. And then, ME-NBI is performed likewise. The final treatment plan is determined by the EUS result, so group assignment does not affect the final treatment plan.

According to clinical stage of early gastric cancer, endoscopic resection is performed in case of endoscopic resection indication or beyond indication but case of having the risk of surgery according to patient status. The surgical resection is performed if the patient wants surgery or does not meet the indications of endoscopic resection.

The pathologist performs a histological evaluation of the resected gastric cancer lesion, including an invasive depth.

B) Study 2 First, the endoscopist performs WLE and describes WLE findings and impression such as location, size, and gross morphology of lesion. The same examiner performs ME-NBI and describes ME-NBI findings and impression such as mucosal pattern, predicted degree of dysplasia.

Endoscopic resection or surgical resection is performed according to the results of histologic result of gastric adenoma.

The pathologist performs a histological evaluation of the resected dysplastic lesion.

ELIGIBILITY:
Inclusion Criteria:

1. Adults over 19 years of age
2. Patients who are diagnosed gastric adenoma or early gastric cancer by esophagogastroduodenoscopy and are planning endoscopic resection or surgical resection for cure.
3. Patients who understand that they have the right to sign the consent form prior to the initiation of treatment and to withdraw from the clinical trial without penalty at any time.

Exclusion Criteria:

1. Failed to obtain informed consent of the patient or guardian.
2. Anyone deemed inappropriate by the researchers or the primary care physician in clinical studies.
3. Women who are pregnant and possibly pregnant or breastfeeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
the accuracy in predicting the invasion depth of EGC. | Within 1 month after lesion resection
  To compare the accuracy of EUS and ME-NBI in predicting the invasion depth of EGC using final pathology result.

SECONDARY OUTCOMES:
The NBI findings that affect the accuracy for predicting of depth. | Within 1 month after lesion resection
  The characteristic imaging findings of ME-NBI for early gastric cancer and gastric adenoma such as microvessels, pits, histological patterns.
  For example) ME-NBI classification Type A : clear regular surface patterns and microvascular architecture. Type B : obscure irregular surface patterns or microvascular architecture. Type C :no surface pattern and sparse microvessels or with avascular areas. Finally, to evaluate the efficacy of ME-NBI for early gastric cancer and gastric adenoma diagnosis.

IPD SHARING:
Plan to Share IPD: No
The information related to this study will be used purely for research purposes and all data will be encrypted and strictly kept confidential and protected. In order to protect the personal information of the patient, information about the patient's identity and information about the patient will be managed as independent data.

REFERENCES:
- [Result] Choi J, Kim SG, Im JP, Kim JS, Jung HC, Song IS. Endoscopic prediction of tumor invasion depth in early gastric cancer. Gastrointest Endosc. 2011 May;73(5):917-27. doi: 10.1016/j.gie.2010.11.053. Epub 2011 Feb 11. PMID 21316050
- [Result] Pei Q, Wang L, Pan J, Ling T, Lv Y, Zou X. Endoscopic ultrasonography for staging depth of invasion in early gastric cancer: A meta-analysis. J Gastroenterol Hepatol. 2015 Nov;30(11):1566-73. doi: 10.1111/jgh.13014. PMID 26094975
- [Result] Kwee RM, Kwee TC. The accuracy of endoscopic ultrasonography in differentiating mucosal from deeper gastric cancer. Am J Gastroenterol. 2008 Jul;103(7):1801-9. doi: 10.1111/j.1572-0241.2008.01923.x. Epub 2008 Jun 28. PMID 18564110
- [Result] Serrano OK, Huang K, Ng N, Yang J, Friedmann P, Libutti SK, Kennedy TJ. Correlation between preoperative endoscopic ultrasound and surgical pathology staging of gastric adenocarcinoma: A single institution retrospective review. J Surg Oncol. 2016 Jan;113(1):42-5. doi: 10.1002/jso.24098. Epub 2016 Jan 19. PMID 26784562
- [Result] Gono K. Narrow Band Imaging: Technology Basis and Research and Development History. Clin Endosc. 2015 Nov;48(6):476-80. doi: 10.5946/ce.2015.48.6.476. Epub 2015 Nov 30. PMID 26668792
- [Result] Hayee B, Inoue H, Sato H, Santi EG, Yoshida A, Onimaru M, Ikeda H, Kudo SE. Magnification narrow-band imaging for the diagnosis of early gastric cancer: a review of the Japanese literature for the Western endoscopist. Gastrointest Endosc. 2013 Sep;78(3):452-61. doi: 10.1016/j.gie.2013.03.1333. Epub 2013 Apr 28. No abstract available. PMID 23632326
- [Result] Kikuchi D, Iizuka T, Hoteya S, Yamada A, Furuhata T, Yamashita S, Domon K, Nakamura M, Matsui A, Mitani T, Ogawa O, Watanabe S, Kaise M. Usefulness of magnifying endoscopy with narrow-band imaging for determining tumor invasion depth in early gastric cancer. Gastroenterol Res Pract. 2013;2013:217695. doi: 10.1155/2013/217695. Epub 2013 Jan 17. PMID 23401676
- [Result] Yagi K, Saka A, Nozawa Y, Nakamura A, Umezu H. Prediction of submucosal gastric cancer by narrow-band imaging magnifying endoscopy. Dig Liver Dis. 2014 Feb;46(2):187-90. doi: 10.1016/j.dld.2013.09.003. Epub 2013 Oct 21. PMID 24157380
- [Result] Jang JY. The Usefulness of Magnifying Endoscopy and Narrow-Band Imaging in Measuring the Depth of Invasion before Endoscopic Submucosal Dissection. Clin Endosc. 2012 Nov;45(4):379-85. doi: 10.5946/ce.2012.45.4.379. Epub 2012 Nov 30. PMID 23251885
- [Result] Kobara H, Mori H, Fujihara S, Kobayashi M, Nishiyama N, Nomura T, Kato K, Ishihara S, Morito T, Mizobuchi K, Iwama H, Masaki T. Prediction of invasion depth for submucosal differentiated gastric cancer by magnifying endoscopy with narrow-band imaging. Oncol Rep. 2012 Sep;28(3):841-7. doi: 10.3892/or.2012.1889. Epub 2012 Jun 26. PMID 22752002
- [Result] Spolverato G, Ejaz A, Kim Y, Squires MH, Poultsides GA, Fields RC, Schmidt C, Weber SM, Votanopoulos K, Maithel SK, Pawlik TM. Use of endoscopic ultrasound in the preoperative staging of gastric cancer: a multi-institutional study of the US gastric cancer collaborative. J Am Coll Surg. 2015 Jan;220(1):48-56. doi: 10.1016/j.jamcollsurg.2014.06.023. Epub 2014 Jul 18. PMID 25283742
- [Result] Li HY, Dai J, Xue HB, Zhao YJ, Chen XY, Gao YJ, Song Y, Ge ZZ, Li XB. Application of magnifying endoscopy with narrow-band imaging in diagnosing gastric lesions: a prospective study. Gastrointest Endosc. 2012 Dec;76(6):1124-32. doi: 10.1016/j.gie.2012.08.015. Epub 2012 Sep 29. PMID 23025977
- [Result] Nonaka T, Inamori M, Honda Y, Kanoshima K, Inoh Y, Matsuura M, Uchiyama S, Sakai E, Higurashi T, Ohkubo H, Iida H, Endo H, Fujita K, Kusakabe A, Atsukawa K, Takahashi H, Tateishi Y, Maeda S, Ohashi K, Nakajima A. Can magnifying endoscopy with narrow-band imaging discriminate between carcinomas and low grade adenomas in gastric superficial elevated lesions? Endosc Int Open. 2016 Nov;4(11):E1203-E1210. doi: 10.1055/s-0042-117632. Epub 2016 Oct 20. PMID 27853747
- [Result] Yoshifuku Y, Sanomura Y, Oka S, Kuroki K, Kurihara M, Mizumoto T, Urabe Y, Hiyama T, Tanaka S, Chayama K. Clinical Usefulness of the VS Classification System Using Magnifying Endoscopy with Blue Laser Imaging for Early Gastric Cancer. Gastroenterol Res Pract. 2017;2017:3649705. doi: 10.1155/2017/3649705. Epub 2017 May 15. PMID 28596787